CLINICAL TRIAL: NCT05359744
Title: A Pilot-study on Multi-level Molecular Profiling of Peak Performance in Endurance Sports
Brief Title: Multi-level Molecular Profiling of Peak Performance in Endurance Sports
Acronym: MSSA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Paracelsus Medical University (Other)
Collaborators: Department of Psychiatry University of Bonn (Other)
Responsible Party: Principal Investigator, Jens Stepan, MD, PhD, Principal Investigator, Paracelsus Medical University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: jestep032022
Record Dates: First submitted 2022-04-25; First posted 2022-05-04 (Actual); Last update posted 2022-05-04 (Actual); Status verified 2022-04

CONDITIONS: Exercise; Exercise Test; Physical Fitness; Healthy
Keywords: Exercise Test; Autophagy; Multi-omic; Fitness level
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Intervention Model Description: 3 groups undergoing intervention, 1 control group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Elite cyclists, male (Experimental): Bicycle ergometer-based exercise testing. 15 min aerobic warm-up phase (2 W/kg) followed by a standardized but individualized ramp-bicycle ergometer protocol to reach maximal exercise capacity after 8 - 12 minutes. The exclusively aerobic energy supply during warm-up will be assessed by constant respiratory quotient and constant arterial lactate concentration (<0.5 mmol in the last 5 min). During exercise, respiratory gas exchange, heart rate, blood pressure, ECG and ratings of perceived exertion will be continuously monitored. Venous blood specimens will be collected before exercise (baseline), at the end of the warm-up as well as 2 min, 10 min, and 30 min in recovery.
  Interventions: Diagnostic Test: Performance testing
- Recreational athletes, male (Experimental): Bicycle ergometer-based exercise testing. 15 min aerobic warm-up phase (1 W/kg) followed by a standardized but individualized ramp-bicycle ergometer protocol to reach maximal exercise capacity after 8 - 12 minutes. The exclusively aerobic energy supply during warm-up will be assessed by constant respiratory quotient and constant arterial lactate concentration (<0.5 mmol in the last 5 min). During exercise, respiratory gas exchange, heart rate, blood pressure, ECG and ratings of perceived exertion will be continuously monitored. Venous blood specimens will be collected before exercise (baseline), at the end of the warm-up as well as 2 min, 10 min, and 30 min in recovery.
  Interventions: Diagnostic Test: Performance testing
- Recreational athletes, female (Experimental): Bicycle ergometer-based exercise testing. 15 min aerobic warm-up phase (1 W/kg) followed by a standardized but individualized ramp-bicycle ergometer protocol to reach maximal exercise capacity after 8 - 12 minutes. The exclusively aerobic energy supply during warm-up will be assessed by constant respiratory quotient and constant arterial lactate concentration (<0.5 mmol in the last 5 min). During exercise, respiratory gas exchange, heart rate, blood pressure, ECG and ratings of perceived exertion will be continuously monitored. Venous blood specimens will be collected before exercise (baseline), at the end of the warm-up as well as 2 min, 10 min, and 30 min in recovery.
  Interventions: Diagnostic Test: Performance testing
- Control, male (No Intervention): Venous blood specimens will be collected at the same time points in the absence of exercise.

INTERVENTIONS:
Diagnostic Test: Performance testing — Performance testing on a bicycle ergometer.
  Arms: Elite cyclists, male; Recreational athletes, female; Recreational athletes, male

SUMMARY:
Physical activity triggers complex molecular responses, including changes in immune-, stress-, and metabolic pathways. For example, autophagy is essential for energy and cellular homeostasis through protein catabolism, and dysregulation results in compromised proteostasis, reduced exercise performance, and excessive secretion of signaling molecules and inflammatory proteins. However, previous research has been limited by the extend of molecules measured and biological processes covered. A better understanding of these processes through multi-omic analysis can improve knowledge of molecular changes in response to exercise. The main purpose of the investigators study is to analyze the effects of acute exercise in correlation to autophagy and other signaling cascades. Specifically, the investigators plan to perform multi-level molecular profiling in a cohort of healthy male elite cyclists and male and female recreational athletes, before, during, and after a bicycle ergometer test. The results will be compared to a control cohort without intervention.

DETAILED DESCRIPTION:
This is a non-randomized controlled trial performed at the Paracelsus Medical University, Salzburg, Austria. The study will recruit 80 healthy men and women. Subjects who meet the inclusion criteria will be allocated to four arms (n = 20 in all groups): 1. elite cyclists, 2. male recreational athletes, 3. female recreational athletes, 4. male control group.

After overnight fasting and medical check-up, groups 1-3 will undergo a bicycle ergometer-based exercise protocol designed to span low (aerobic) to severe (anaerobic) domains of exercise. The protocol consists of a 15 min aerobic warm-up phase followed by a ramp-bicycle ergometer protocol.

During exercise, performance-relevant data will be continuously monitored. Venous blood specimens will be collected before exercise (baseline), at the end of the warm-up as well as 2 min, 10 min, and 30 min in recovery.

ELIGIBILITY:
Inclusion Criteria:

* All arms: ability to give written informed consent
* Arms 1- 3: inconspicuous medical examination (medical history, resting ECG, echocardiography)
* Elite athletes (arm1, cyclists): maximum oxygen uptake > 65 ml/kg/KG
* Elite athletes (arm1, cyclists): participation in cycling competitions on a regular basis
* Recreational athletes (arms 2 and 3): maximum oxygen uptake < 65 ml/kg/KG for male subjects and < 55 ml/kg/KG for female subjects

Exclusion Criteria:

* All arms: unable to communicate adequately by language
* All arms: regular use of prescription drugs other than thyroxine or antihistamines
* All arms: alcohol consumption as equivalent doses averaging more than 40 g of pure alcohol per day
* All arms: use of illicit drugs
* All arms: known diseases of the cardiovascular system
* All arms: arterial hypertension over 160/90 mmHg at rest
* All arms: known pulmonary diseases, especially bronchial asthma
* All arms: surgery less than 4-6 months ago.
* All arms: abnormalities in the medical examination (medical history, resting ECG, echocardiography)
* Arms 1-3: orthopaedic diseases that preclude maximum exercise on a bicycle ergometer
* Elite athletes (arm1, cyclists): maximum oxygen uptake < 65 ml/kg/KG
* Recreational athletes (arms 2 and 3): maximum oxygen uptake > 65 ml/kg/KG for male subjects and > 55 ml/kg/KG for female subjects
* Arm 3: positive urine ß-HCG

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2021-10-15 (Actual); Primary Completion 2022-10-15 (Estimated); Study Completion 2022-10-15 (Estimated)

PRIMARY OUTCOMES:
Proteomics and autophagy processes | Before the exercise test (baseline), at the end of the 15 minute warm-up phase and 2 minutes, 10 minutes and 30 minutes after termination of the exercise test.
  Change in protein levels of autophagy biomarkers (LC3II & p62) of isolated PBMCs (peripheral blood mononuclear cells) by Western Blotting.

SECONDARY OUTCOMES:
Salivary cortisol levels | Before the exercise test (baseline), at the end of the 15 minute warm-up phase and 2 minutes, 10 minutes and 30 minutes after termination of the exercise test.
  Salivary cortisol levels in nmol per Liter (nmol/L) after will be evaluated and compared to the control group
Proteome patterns | Before the exercise test (baseline), at the end of the 15 minute warm-up phase and 2 minutes, 10 minutes and 30 minutes after termination of the exercise test.
  Change in protein levels and protein phosphorylation by untargeted mass spectrometry-based proteomics and phosphoproteomics of isolated PBMCs (peripheral blood mononuclear cells).
Metabolic processes | Before the exercise test (baseline), at the end of the 15 minute warm-up phase and 2 minutes, 10 minutes and 30 minutes after termination of the exercise test.
  Targeted and quantitative analysis by mass spectrometry of change in metabolites of Plasma.
Lipid profiling | Before the exercise test (baseline), at the end of the 15 minute warm-up phase and 2 minutes, 10 minutes and 30 minutes after termination of the exercise test.
  Targeted and quantitative analysis by mass spectrometry of change in plasma Lipids.
Phosphoproteome patterns | Before the exercise test (baseline), at the end of the 15 minute warm-up phase and 2 minutes, 10 minutes and 30 minutes after termination of the exercise test.
  Change in protein phosphorylation by untargeted mass spectrometry-based phosphoproteomics of isolated PBMCs (peripheral blood mononuclear cells).
Ubiquitinome patterns | Before the exercise test (baseline), at the end of the 15 minute warm-up phase and 2 minutes, 10 minutes and 30 minutes after termination of the exercise test.
  Change in protein ubiquitination levels by untargeted mass spectrometry-based proteomics of isolated PBMCs (peripheral blood mononuclear cells).
Epigenetic patterns | Before the exercise test (baseline), at the end of the 15 minute warm-up phase and 2 minutes, 10 minutes and 30 minutes after termination of the exercise test.
  Evaluate epigentic methylation patterns through blood based epigenome analysis
Exosomal protein patterns | Before the exercise test (baseline), at the end of the 15 minute warm-up phase and 2 minutes, 10 minutes and 30 minutes after termination of the exercise test.
  Evaluate exosomal protein content through mass spectrometry based analysis

CONTACTS AND LOCATIONS:
Overall Officials: Jens Stepan, MD, PhD, Principal Investigator — Department of Obstetrics and Gynecology, University Hospital Salzburg, Austria
Locations (1):
- Paracelsus Medical University, Salzburg, Austria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Hasin Y, Seldin M, Lusis A. Multi-omics approaches to disease. Genome Biol. 2017 May 5;18(1):83. doi: 10.1186/s13059-017-1215-1. PMID 28476144
- [Result] Nicora G, Vitali F, Dagliati A, Geifman N, Bellazzi R. Integrated Multi-Omics Analyses in Oncology: A Review of Machine Learning Methods and Tools. Front Oncol. 2020 Jun 30;10:1030. doi: 10.3389/fonc.2020.01030. eCollection 2020. PMID 32695678
- [Result] Contrepois K, Wu S, Moneghetti KJ, Hornburg D, Ahadi S, Tsai MS, Metwally AA, Wei E, Lee-McMullen B, Quijada JV, Chen S, Christle JW, Ellenberger M, Balliu B, Taylor S, Durrant MG, Knowles DA, Choudhry H, Ashland M, Bahmani A, Enslen B, Amsallem M, Kobayashi Y, Avina M, Perelman D, Schussler-Fiorenza Rose SM, Zhou W, Ashley EA, Montgomery SB, Chaib H, Haddad F, Snyder MP. Molecular Choreography of Acute Exercise. Cell. 2020 May 28;181(5):1112-1130.e16. doi: 10.1016/j.cell.2020.04.043. PMID 32470399
- [Result] Mukherjee K, Edgett BA, Burrows HW, Castro C, Griffin JL, Schwertani AG, Gurd BJ, Funk CD. Whole blood transcriptomics and urinary metabolomics to define adaptive biochemical pathways of high-intensity exercise in 50-60 year old masters athletes. PLoS One. 2014 Mar 18;9(3):e92031. doi: 10.1371/journal.pone.0092031. eCollection 2014. PMID 24643011
- [Result] De Pauw K, Roelands B, Cheung SS, de Geus B, Rietjens G, Meeusen R. Guidelines to classify subject groups in sport-science research. Int J Sports Physiol Perform. 2013 Mar;8(2):111-22. doi: 10.1123/ijspp.8.2.111. PMID 23428482
- [Result] Martin DT, McLean B, Trewin C, Lee H, Victor J, Hahn AG. Physiological characteristics of nationally competitive female road cyclists and demands of competition. Sports Med. 2001;31(7):469-77. doi: 10.2165/00007256-200131070-00002. PMID 11428684
- [Result] Hoffman NJ. Omics and Exercise: Global Approaches for Mapping Exercise Biological Networks. Cold Spring Harb Perspect Med. 2017 Oct 3;7(10):a029884. doi: 10.1101/cshperspect.a029884. PMID 28348175